CLINICAL TRIAL: NCT04585139
Title: Assessing Non-adjunctive CGM Safety at Home and in New Markets
Acronym: ANSHIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PTL-903833
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study consists of two phases. Phase I is a single-arm, prospective, multicenter, interventional design. Phase II is a randomized controlled arm study during which participants will be randomized 1:1 to Commercial CGM or Updated CGM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Phase 1 -- Introduction to Dexcom G6 CGM (Other): A 2 week run-in wear period of blinded CGM followed by 12 weeks of wear of a Commercially available CGM
  Interventions: Device: Phase 1- Introduction to Dexcom G6 CGM
- Phase 2 -- Comparison of an Updated G6 Transmitter to Commercial Dexcom G6 CGM (Active Comparator): 1 group will wear a Commercially available CGM for 12 weeks while the 2 group will wear an Updated CGM for 12 weeks.
  Interventions: Device: Phase 1- Introduction to Dexcom G6 CGM

INTERVENTIONS:
Device: Phase 1- Introduction to Dexcom G6 CGM — Examine whether non-adjunctive use of CGM improves glycemic control in adults with diabetes managed by intensive insulin therapy

SUMMARY:
The purpose of the study is to examine whether non-adjunctive (without having to double check using another method) use of Continuous Glucose Monitoring improves A1c in adults or children with diabetes managed by intensive insulin therapy.

ELIGIBILITY:
Inclusion Criteria

* Age 2 years or older
* A diagnosis of T1D or T2D made at least 6 months prior to enrollment. At least 20 adult participants will have T1D; and 10 will have T2D; 10 participants will be over age 65 years.
* Using IIT (either an insulin pump or MDI)
* HbA1c value ≥ 7.5% (≥ 58 mmol/mol) measured by local lab within prior 30-days before enrollment or by point of care at time of screening.
* eGFR ≥ 30 within the last 90-days prior to enrollment (adult participants only)
* Currently performing 2 or more SMBG fingersticks a day by historical average and willing to continue this during the blinded CGM wear.

Exclusion Criteria

* Use of real-time or intermittently scanned CGM in the 6 months prior to enrollment.
* BMI > 45.
* Anticipated changes to insulin delivery method or insulin formulation(s).
* Insulin formulation changes within class will be permitted if required per formulary change and represent equivalent therapy (eg: insulin lispro change to insulin aspart).
* Pregnancy (as demonstrated by a positive test at study entry) at time of screening or are planning to become pregnant during the study.
* Applicable only to women of reproductive potential.
* Planned or currently using weight reduction medications, programs or surgery. Defined as 1) using weight loss medications and losing weight (e.g. chronic use of weight loss medications with stable weight is not exclusionary) or planning on using weight loss prescription medication during the study; 2) currently using or planning on initiating a modified fasting program (e.g. protein-sparing diet plans) during the study; or 3) bariatric surgical procedure within the past year or plans for undergoing bariatric surgery during the study.
* Concomitant disease or condition that may compromise patient safety including, but not limited to; severe mental illness, a diagnosed or suspected eating disorder or any uncontrolled long-term medical/psychiatric condition that would interfere with study- related tasks or visits, including ongoing treatment for a significant malignancy. These assessments/conditions are made at investigator's discretion.
* Known (or suspected) significant allergy to medical-grade adhesives.
* Any condition, per investigator assessment, that could impact the stability of the HbA1c measurement, for example,
* Acute or chronic blood loss or bleeding disorder,
* Red blood cell transfusion or erythropoietin, administration in the 3 months prior to enrollment,
* Or red blood cell transfusion or erythropoietin administration anticipated during the course of the study.
* Anticipated acute use of oral or injectable glucocorticoids that could affect glycemic control and impact HbA1c, for example,
* Frequent steroid bursts used for inflammatory arthritis or inflammatory bowel disease,
* Or recurrent lumbar epidural steroid injections,
* Current treatment with hydroxyurea
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  Phase 1 change in HbA1c for the adult cohort only.

CONTACTS AND LOCATIONS:
Locations (1):
- Las Vegas Endocrinology, Henderson, Nevada, United States

IPD SHARING:
Plan to Share IPD: No